CLINICAL TRIAL: NCT05486416
Title: A Global Multicenter, Randomized, Double-blinded, Propofol-controlled, Phase 3 Clinical Study to Evaluate the Efficacy and Safety of HSK3486 Injectable Emulsion for Induction of General Anesthesia in Adults Undergoing Elective Surgery
Brief Title: Safety and Efficacy of HSK3486 Compared to Propofol for Induction of General Anesthesia in Adults With Elective Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco-USA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK3486-309
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: General Anesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Intervention Model Description: Surgical pre-induction analgesia
Who Masked: Participant
Masking Description: Double blinded, 2:1 ratio of HSK3489 and Propofol respectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HSK3486 for general anesthesia induction (Experimental): HSK3486 for induction of general anesthesia
  Interventions: Drug: HSK3486
- Propofol for general anesthesia induction (Active Comparator): Propofol for induction of general anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — HSK3486 for induction of general anesthesia
  Arms: HSK3486 for general anesthesia induction
Drug: Propofol — Propofol for induction of general anesthesia
  Other Names: Diprivan
  Arms: Propofol for general anesthesia induction

SUMMARY:
To demonstrate HSK3486 0.4/0.2 mg/kg (0.4 mg/kg intravenous [IV] slow injection over 30 [±5] seconds for the first dose, an additional 0.2 mg/kg if needed) is non-inferior to Propofol 2.0/1.0 mg/kg (2.0 mg/kg IV slow injection over 30 [±5] seconds for first dose, an additional 1.0 mg/kg if needed) in success of induction of general anesthesia in adults undergoing elective surgery.

DETAILED DESCRIPTION:
This is a global multicenter, randomized, double-blinded, propofol-controlled, phase 3 clinical study to evaluate the efficacy and safety of HSK3486 for induction of general anesthesia in adults undergoing elective surgery with endotracheal intubation.

After screening, eligible subjects will be randomized in a 2:1 ratio to receive either HSK3486 0.4/0.2 mg/kg (i.e., 0.4 mg/kg IV slow injection over 30 [±5] seconds followed by an additional 0.2 mg/kg dose over 10 [±2] seconds if needed) or propofol 2.0/1.0 mg/kg (i.e., 2.0 mg/kg IV slow injection over 30 [±5] seconds followed by an additional 1.0 mg/kg dose over 10 [±2]seconds if needed) in a blinded manner. Enrolled subjects will be stratified by American Society of Anesthesiologists Physical Status (ASA-PS; I-II and III-IV), age (<65 and ≥65 years), and Body Mass Index (BMI <35 and ≥35 kg/m2). Endotracheal intubation will be performed after adequate anesthetic induction (Modified Observer's Assessment of Awareness/Sedation [MOAA/S] ≤1) (Appendix 1) has been achieved and administration of neuromuscular blocking agent.

Before surgery, premedication is allowed except for sedative-hypnotic or analgesic drugs. Premedication should be recorded if used.

Prior to administration of the study drug in the operating room, the preoperative readiness of each subject will be confirmed. Oxygen will be supplied through a facemask (oxygen flow rate: ≥4 L/min) at least 2 minutes before study drug administration. Subsequently, the investigator can adjust the oxygen flow according to the specific situation of the subject and maintenance IV solution (normal saline [NS], lactated ringer's [LR], or 5% dextrose) will be administrated through IV infusion. Throughout the pre-induction and induction periods, a timing device must be used to allow accuracy and sequencing of necessary assessments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy all of the following criteria at the screening visit:

  1. Subjects undergoing elective surgery (non-emergency, non-cardiothoracic, and non-intracranial surgery anticipated to last at least 1 hour) requiring endotracheal intubation and inhalation general anesthesia during the maintenance period. Duration of surgery is defined as time from study drug administration to time of transfer from operating room to recovery room or PACU.
  2. Males or females, aged ≥18 years old, with ASA PS I to IV (Appendix 6). For ASA-PS IV subjects, clinical status must be optimized at time of preoperative anesthesia evaluation per judgement of the anesthesiologist.
  3. BMI ≥18 kg/m2.
  4. Vital signs at screening: RR ≥10 and ≤24 breaths/min; SpO2 ≥92% in ambient air; SBP ≥90 and ≤160 mmHg; DBP ≥55 and ≤ 100 mmHg; HR ≥55 (or ≥50 if subjects are on beta blockers) and ≤100 beats/min.
  5. For all women of childbearing potential, negative serum pregnancy test within the screening period and negative urine pregnancy test at baseline (Day 1). Additionally, women of childbearing potential* and male subjects with female partners of childbearing potential must agree to use contraception as defined in 7.3.4 from the time of consent until 30 days post study drug administration.
  6. For subjects with known hypothyroidism and/or on thyroid-hormone replacement treatment (i.e., thyroxine), or subjects suspected to have thyroid dysfunction based on clinical laboratory and physical exam, a TSH must drawn and be within normal levels.
  7. Capable of understanding the procedures and methods of this study, willing to sign an Informed Consent Form (ICF), and able to complete this study in strict compliance with the study protocol.
  8. Willing to comply with the site's COVID guidelines and testing requirements as applicable.
  9. Patients with psychiatric/mental disorders must be considered stable on treatment (e.g., SSRIs, SNRIs, TCAs, MAOIs, psychotherapy) per investigator judgement, and no hospitalizations and urgent care due to the underlying psychiatric pathology for at least 12 months.

     * Women are considered of childbearing potential until becoming post-menopausal, unless she had a documented hysterectomy or bilateral oophorectomy / salpingo-oophorectomy. A woman is considered to be post-menopausal if she had no menses for at least 12 consecutive months (without an alternative medical cause).

Exclusion Criteria:

1. Contraindications to deep sedation/general anesthesia or a history of adverse reaction to sedation/general anesthesia.
2. Known to be allergic to eggs, soy products, opioids and their antidotes, or propofol; subjects having contraindications to propofol, opioids, and their antidotes. In cases where the only previous reaction to opioids was itching or nausea, subjects need not be excluded if the investigator believes the subject is not truly allergic to opioids.
3. Medical condition or evidence of increased sedation/general anesthesia risk as follows:

   1. Cardiovascular disorder: uncontrolled hypertension (SBP >160 mmHg and/or DBP >100 mmHg) with or without antihypertensive therapy (antihypertensive therapy should be stable for 1 month prior to screening), serious arrhythmia (including the subjects with implanted pace makers), unstable heart failure, Adams-Stokes syndrome (i.e., syncope or near-syncope due to cardiac arrythmia), unstable angina, myocardial infarction occurring within 6 months prior to screening, history of tachycardia/bradycardia requiring medications, third degree atrioventricular block or QT interval corrected for HR using Fridericia's formula (QTcF) ≥450 ms for males and ≥470 ms for females.
   2. History of severe obstructive lung disease (i.e., forced expiratory volume in 1 second [FEV1] <50% predicted), history of bronchospasm requiring treatment in a hospital emergency room or hospitalization occurring within 3 months prior to screening, developing acute respiratory tract infection within 2 weeks prior to baseline (such as symptoms of fever, shortness of breath, wheezing, nasal congestion, and cough).
   3. Cerebrovascular disease: subject with a history of serious craniocerebral injury, convulsion, seizure disorder, intracranial hypertension, cerebral aneurysm, or stroke.
   4. Patients with psychiatric/mental disorders who have not been on a stable treatment regimen (e.g., SSRIs, SNRIs, TCAs, MAOIs, psychotherapy) per investigator judgement, for at least 12 months or who have been hospitalized or had emergent/urgent care due to the underlying psychiatric pathology within the last 12 months.
   5. Uncontrolled clinically significant conditions of liver (e.g., severe hepatic insufficiency defined as Childs-Pugh class C), kidney, gastrointestinal tract, blood system, nervous system, or metabolic system diseases, judged by the investigator to be unsuitable for involvement in the study.
   6. History of uncontrolled diabetes in the opinion of the investigator.
   7. History of alcohol abuse within 3 months prior to screening, where alcohol abuse refers to daily alcohol drinking >2 units of alcohol (1 unit = 360 mL of beer or 45 mL of spirit with a strength of 40% or 150 mL of wine).
   8. History of drug abuse that, in the opinion of the investigator, may confound the interpretation of safety or efficacy in a study subject.
   9. For subjects with known hypothyroidism and/or on thyroid-hormone replacement treatment (i.e., thyroxine), or subjects suspected to have thyroid dysfunction based on clinical laboratory and physical exam who has a TSH value outside the normal range.
4. Management risks of respiratory tract and judged by the investigator to be unsuitable for inclusion in the study as follows:

   1. Asthma must be stable: stable doses of asthma medications for the past 6 months, no requirement for rescue inhalers or oral steroids within past 6 months, not evaluated in emergency department, urgent care, or hospitalized for an asthma attack within past 1 year.
   2. History (or family history) of malignant hyperthermia.
   3. Any previous failure of tracheal intubation.
   4. Judged to have a difficult airway for endotracheal intubation in the opinion of the Investigator based on parameters such as modified Mallampati score (Grade III or IV [Appendix 7]), neck mobility, short thyromental distance, and/or history of difficult intubation).
5. Any medication that has the potential to interact synergistically with propofol or HSK3486, including but not limited to all sedatives and hypnotics (e.g., benzodiazepines and opioids), taken within 5 half-lives prior to Day 1.
6. Laboratory parameters measured at screening with the following levels:

   1. Neutrophil count ≤1.5 x 109/L
   2. Platelet count <80 x 109/L
   3. Hemoglobin <90 g/L (without blood transfusion within 14 days)
   4. Alanine transaminase and/or aspartate transaminase ≥2.0 x upper limit of normal (ULN)
   5. Total bilirubin ≥2.0 x ULN
   6. Severe renal impairment defined by creatinine clearance (CrCl) ≤30 mL/min
7. Female subjects with a positive pregnancy test at screening (serum) or baseline (urine); lactating subjects; any subject planning to get pregnant within 1 month after the study (including the male subject's partner).
8. Judged by the investigator to have any other factors that make the subject unsuitable for participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (21):
  - North Alabama Medical Center, Florence, Alabama
  - Helen Keller Hospital, Sheffield, Alabama
  - University of Miami Hospital, Miami, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - EBGS Clinical Research Center, Snellville, Georgia
  - University of Iowa Hospitals and Clinics (Dept of Anesthesia), Iowa City, Iowa
  - U of L Health, University of Louisville Hospital, Louisville, Kentucky
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - M3-Emerging Medical Research, LLC, Durham, North Carolina
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - The Ohio State University Wexner Medical Center - University Hospital, Columbus, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Village, Houston, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Endeavor Clinical Trials, LLC, San Antonio, Texas
- Poland (3):
  - Uniwersytecki Szpital Kliniczny W Opolu, Opole
  - Państwowy Instytut Medyczny Mswia - Klinika Anestezjologii I Intensywnej Terapii, Warsaw
  - Spsk Nr 1 Im. Prof. S. Szyszko, Zabrze
- Spain (4):
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital General Universitario De Ciudad Real, Ciudad Real
  - Universidad de Navarra - Clinica Universidad de Navarra en Pamplona, Pamplona
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- HSK3486: HSK3486 for general anesthesia induction
  HSK3486: HSK3486 for induction of general anesthesia
- Propofol: Propofol for general anesthesia induction
  Propofol: Propofol for induction of general anesthesia.
Period: Overall Study
Arm/Group | HSK3486 | Propofol
Started | 313 | 152
Dosed | 300 | 145
Full Analysis Set | 300 | 145
Safety Set | 300 | 145
Completed | 300 (completed primary efficacy measurement) | 145 (completed primary efficacy measurement)
Not Completed | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSK3486 for General Anesthesia Induction | Propofol for General Anesthesia Induction | Total
Number analyzed (Participants) | 300 | 145 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 229 | 110 | 339
  >=65 years | 71 | 35 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 74 | 247
  Male | 127 | 71 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 38 | 129
  Not Hispanic or Latino | 204 | 107 | 311
  Unknown or Not Reported | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 23 | 61
  White | 254 | 114 | 368
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 234 | 119 | 353
  Poland | 27 | 15 | 42
  Spain | 39 | 11 | 50
ASA-PS [Count of Participants; unit: Participants] — ASA-PS is completed preoperatively per judgement of the anesthesiologist:
  ASA I: Normal and healthy. No systemic diseases other than local lesions. ASA II: A subject with mild systemic disease. ASA III: A subject with severe systemic disease that results in functional limitations but not incapacity.
  ASA IV: A subject with severe systemic disease that is a constant threat to life and results in incapacity.
  ASA V: A moribund subject who is not expected to survive without the operation.
  Participants
    ASA-PS I | 47 | 24 | 71
    ASA-PS II | 183 | 90 | 273
    ASA-PS III | 70 | 31 | 101
BMI [Count of Participants; unit: Participants]
  <35kg/m^2 | 237 | 113 | 350
  ≥35kg/m^2 | 63 | 32 | 95

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of General Anesthesia Induction
Description: 1. Induction success (MOAA/S ≤1) after administration of the study drug, and
  2. One or less top-up doses required without using any rescue drugs.
Time Frame: From the time of study drug administration to desired depth of anesthesia to MOAA/S≤1( up to 5 minutes)
Population: Completed primary efficacy measurement
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 300 | 145
Participants | 298 | 143

2. Secondary Outcome: Percentage of Subjects With Successful Induction Who Maintain the Desired Depth of Anesthesia for General Elective Surgery, AND Without Significant Cardiac and Respiratory Depression
Description: The outcome is defined by all the following conditions:
  a) Desired depth of anesthesia for general elective surgery is defined if all following criteria are met: i) No clinical signs of inadequate depth of anesthesia, such as lacrimation, movement, vomiting, coughing, laryngospasm, bucking, swallowing reflex or bronchospasm etc.
  ii) No blood pressure (SBP, DBP, or MAP) increases more than 20% from baseline in response to any major operational procedures or noxious stimulus in defined period.
  iii) Subjects maintain desired depth of anesthesia for general elective surgery with BIS as an objective assessment (after reaching initial lowest value, BIS remains sustainable level at not more than 60).
  b) No significant respiratory depression, such as apnea, prior to the administration of rocuronium bromide.
  c) No significant cardiac depression indicated by blood pressure decrease that requires intervention, i.e., vasopressors and/or IV fluid resuscitation.
Time Frame: 15 minutes from end of drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 for General Anesthesia Induction | Propofol for General Anesthesia Induction
Number analyzed (Participants) | 300 | 145
Participants | 81 | 45

3. Secondary Outcome: Proportion of Subjects With Any Injection-site Pain on Numeric Rating Scale ≥1
Description: 0 = No Pain 1-3 = Mild Pain 4-6 = Moderate Pain 7-9 = Severe Pain 10 = Worst pain imaginable
Time Frame: From start of the drug administration to MOAA/S ≤1 (up to 3 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 for General Anesthesia Induction | Propofol for General Anesthesia Induction
Number analyzed (Participants) | 300 | 145
Participants | 56 | 86

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time of informed consent until the final study visit (Day 8). A treatment-emergent AE is defined as: an AE that occurs after the subject starts treatment with the IMP. If an Investigator becomes aware of a serious adverse event within 30 days after the last dose of study drug and it is considered by him/her to be caused by the study drug with a reasonable possibility, the event must be documented and reported.
Description: Adverse Events of Special Interest (AESIs) due to pharmacological effect of an anesthetic agent include hypoxemia, bradycardia, severe hypotension, allergy/anaphylaxis, cardiac arrhythmia and QTc prolongation.
Arm/Group | HSK3486 for General Anesthesia Induction | Propofol for General Anesthesia Induction
All-Cause Mortality (participants affected / at risk) | 1/300 | 0/145
Serious Adverse Events (participants affected / at risk) | 5/300 | 1/145
Other Adverse Events (participants affected / at risk) | 185/300 | 96/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSK3486 for General Anesthesia Induction (N=300) | Propofol for General Anesthesia Induction (N=145)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Mediastinal hematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urecteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Internal hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Wound dehiscence (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HSK3486 for General Anesthesia Induction (N=300) | Propofol for General Anesthesia Induction (N=145)
Hypotension (Vascular disorders) | 55 | 32
Hypertension (Vascular disorders) | 24 | 9
Procedural Hypotension (Injury, poisoning and procedural complications) | 34 | 23
Procedural Pain (Injury, poisoning and procedural complications) | 9 | 6
Procedural nausea (Injury, poisoning and procedural complications) | 4 | 5
Nausea (Gastrointestinal disorders) | 48 | 17
Constipation (Nervous system disorders) | 3 | 10
Tachycardia (Cardiac disorders) | 13 | 7
Electrocardiogram QT prolonged (Investigations) | 2 | 5
Haematuria (Renal and urinary disorders) | 4 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: HSK3486-309 Protocol V9.0 (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT05486416/Prot_SAP_000.pdf
  • Statistical Analysis Plan: HSK3486-309 Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05486416/SAP_001.pdf